CLINICAL TRIAL: NCT01436019
Title: Analysis of Anti-infliximab, Anti-adalimumab and Anti-etanercept Antibodies in Children and Young Adolescents With Juvenile Idiopathic Arthritis
Brief Title: Study of Antibodies to Anti-TNF Agents in Juvenile Idiopathic Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Blood Transfusion Centre of Slovenia (Other Government)
Collaborators: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Miha Kosmac, dr., Blood Transfusion Centre of Slovenia
Other Study IDs: BTC-PK-1
Record Dates: First submitted 2011-09-13; First posted 2011-09-19 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Juvenile idiopathic arthritis; Rheumatic diseases; Antibodies; Biological therapy
MeSH Terms: conditions — Arthritis, Juvenile; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- anti-TNF treatment: Children or young adolescents with juvenile idiopathic arthritis receiving either infliximab, adalimumab or etanercept.

SUMMARY:
The purpose of this study is to analyze the frequency of the formation of antibodies against three different anti-TNF biologic agents used for the therapy of juvenile idiopathic arthritis.

DETAILED DESCRIPTION:
Juvenile idiopathic arthritis (JIA) is the umbrella term for a heterogeneous group of inflammatory arthropathies that can affect children and young adults and is the most common rheumatic disease of the pediatric population. In high-income countries it has a yearly incidence of 2-20 cases per 100 000 population and a prevalence of 16-150 cases per 100 000 population. Treatment of JIA includes a combination of pharmacological interventions, physical and occupational therapy, and psychosocial support. Although a definitive cure is still not available, the prognosis for patients with JIA has improved greatly in recent years due to improved disease management and with the introduction of biologics that can provide an efficient alternative for patients who are nonresponsive to other treatments. Traditionally, biologic treatments in JIA have focused on blocking one of the central mediators of the inflammatory response, the cytokine tumor necrosis factor (TNF). Currently there are three anti-TNF agents available for the treatment of JIA: infliximab, adalimumab and etanercept. One of the major drawbacks of these therapeutics is the production of anti-drug antibodies (ADA) that have been correlated with an increased risk of adverse events and loss of drug efficacy. The study will evaluate the frequency of the formation of anti-infliximab antibodies in patients treated with infliximab, anti-adalimumab antibodies in patients treated with adalimumab and anti-etanercept antibodies in patients treated with etanercept. A common practice in cases nonresponsive to one of the described anti-TNF agents is the discontinuation of therapy and switching to a different ant-TNF agent. Therefore, the frequency of the formation of antibodies to each of the described anti-TNF agents will also be compared between patients who have previously received a different anti-TNF agent and patients who have not received any previous anti-TNF therapy. The results of this study will highlight the risks of formation of antibodies to three different anti-TNF biologic agents used for the therapy of JIA either alone or after the previous discontinuation of a different anti-TNF agent.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of juvenile idiopathic arthritis
* Must be treated either with infliximab, adalimumab or etanercept

Exclusion Criteria:

* Contraindications to anti-TNF therapy
* Concurrent treatment with any biologic agent other than infliximab, etanercept, or adalimumab
* Previous treatment with rituximab

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Determination of the presence and quantification of anti-drug antibodies by ELISA or other immunoassay. | Up to one year
  In patients receiving infliximab anti-infliximab antibodies will be measured, in patients receiving adalimumab anti-adalimumab antibodies will be measured and in patients receving etanercept anti-etanercept antibodies will be measured. In all cases the primary outcome measure will be the determination of the presence of these antibodies (YES/NO) and their quantification (in EqU compared to a reference serum) using ELISA or other suitable immunoassay.

SECONDARY OUTCOMES:
Determination of the presence and quantification of the serum level of the anti-TNF agent used for JIA therapy by ELISA or other immunoassay. | Up to one year
  In patients receiving infliximab the trough serum level of infliximab will be measured, in patients receiving adalimumab the trough serum level of adalimumab will be measured and in patients receiving etanercept the trough serum level of etanercept will be measured by ELISA or other suitable immunoassay.
Determination of the presence and quantification of the isotypes and subtypes of the anti-drug antibodies by ELISA or other immunoassay. | Up to one year.
  In samples where the presence of anti-infliximab, anti-adalimumab or anti-etanercept antibodies will be confirmed, the isotypes and/or subtypes of the antibodies will be determined by ELISA or other suitable immunoassay.
Time to first detection of anti-drug antibodies. | Up to one year.
  The elapsed time from start of therapy until first detection of anti-drug antibodies will assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Miha Kosmač, PhD, Principal Investigator — Blood Transfusion Centre of Slovenia; Tadej Avčin, MD, PhD, Study Director — University Medical Centre, Ljubljana, Slovenia; Vladka Čurin Šerbec, PhD, Study Chair — Blood Transfusion Centre of Slovenia
Locations (1):
- University Medical Centre, Ljubljana, Slovenia

REFERENCES:
- [Background] Kosmac M, Avcin T, Toplak N, Simonini G, Cimaz R, Curin Serbec V. Exploring the binding sites of anti-infliximab antibodies in pediatric patients with rheumatic diseases treated with infliximab. Pediatr Res. 2011 Mar;69(3):243-8. doi: 10.1203/PDR.0b013e318208451d. PMID 21131896